CLINICAL TRIAL: NCT03661060
Title: BLITZ Heart Failure
Acronym: BLITZ-HF
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K15
Record Dates: First submitted 2018-08-16; First posted 2018-09-07 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
Keywords: Acute Heart Failure; Chronic Heart Failure; Guideline adherence; Clinical registry
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate if Italian Cardiologists are treating Heart Failure (HF) patients according to International guidelines and if a structured educational program can improved their adherence.

DETAILED DESCRIPTION:
Multicentre, cross-sectional, prospective, non-interventional, observational study designed to evaluate the level of adherence to current ESC guidelines recommendations in both acute and chronic HF patients enrolled in each participating center and to verify if a specific HF educational intervention composed by an educational web based program of data collection and face to face meetings is able to improve adherence to guidelines recommendations evaluated during a second enrollment period.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with chronic HF and those admitted for acute (de novo) or worsening chronic HF.
* Chronic HF: any NYHA class (I-IV).
* Acute HF Only patients in NYHA class III or IV, or with pulmonary edema or cardiogenic shock for whom an IV therapy specific for HF (diuretic, vasodilators, vasopressors) is administered.
* Any gender.
* Any etiology of HF.
* Any level of EF.
* Written informed consent.

Exclusion Criteria:

* - Age <18 years.
* Inclusion in registries or trials that can influence, by protocol, the clinical management of patients.
* Patients already enrolled in the BLITZ HF (by another participating centre or in the first enrollment period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized and ambulatory heart failure patients admitted to or evaluated in Italian Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 7569 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Adherence to current guideline | Enrollment
  To assess number of patients managed and treated following the 2016 ESC Heart Failure Gudelines (acute HF, chronic HFrEF, chronic HFmrEF, chronic HFpEF).
Patients managed and treated following International Guideline | 24 months
  Patients treatment in phase 1 versus phase 3

SECONDARY OUTCOMES:
Mortality | 12 months Follow-up
  Death from all-causes, for cardiovascular causes, for HF
Morbidity | 12 months Follow-up
  Hospital admissions from all-causes, for cardiovascular causes, for HF
Indication to heart failure device implantation | Enrollement
  The rate of patients with chronic HFrEF with an indication to ICD and/or CRT planned in clinical practice
Prescription rate of disease modifying drugs | Enrollment
  The rate of patients with HFrEF receiving all the drugs recommended by current guidelines: ACE-Is/ARBs, betablockers and MRAs, in the absence of specific contraindications/intolerance.
Oral anticoagulation prescription in patients with AF | Enrollment
  Rate of patients treated with oral anticoagulants in case of AF
Use of ARNI | Enrollment
  The rate of implementation of a new drug approach (ARNI) for patients with HF and EF ≤35%
Creatinine and EF evaluation | Enrollment
  The rate of CHF patients with an available measure of EF and of creatinine.

CONTACTS AND LOCATIONS:
Locations (123):
- Italy (123):
  - Ospedali Riuniti - Sod Cardiologia Ospedaliera Emod. E Utic, Ancona, AN
  - Ospedale Generale Regionale-Po U. Parini - U.O. Cardiologia E Cure Intensive Card., Aosta, AO
  - Ospedale Gen.Le Prov.Le C.G. Mazzoni - Sc Cardiologia, Ascoli Piceno, AP
  - Ospedale Valdichiana Santa Margherita - Uos Cardiologia E Hdu, Cortona, AR
  - Aorn San Giuseppe Moscati - U.O. Cardiologia/Utic 'D. Rotiroti', Avellino, AV
  - Asst Papa Giovanni Xxiii - Cardiologia 1, Bergamo, BG
  - Ospedale Bolognini - Cardiologia E Unita' Coronarica, Seriate, BG
  - Ospedali Treviglio-Caravaggio - Cardiologia, Treviglio, BG
  - Ospedale Santa Maria Del Prato - U.O. Di Cardiologia, Feltre, BL
  - Ospedale Maggiore - U.O. Di Cardiologia, Bologna, BO
  - Ospedale Policlinico S. Orsola-Malpighi - Medicina Interna - Borghi, Bologna, BO
  - Ospedale Bellaria - U.O. Di Cardiologia, Bologna, BO
  - Ospedale Perrino - U.O.C. Di Cardiologia, Brindisi, BR
  - Spedali Civili - Cardiologia, Brescia, BS
  - Istituto Osped. Fondazione Poliambulanza - Unita' Operativa Di Cardiologia, Brescia, BS
  - Ospedale Civile 'La Memoria' - U.O. Di Cardiologia, Gavardo, BS
  - Ics Maugeri Spa Societa' Benefit - U.O. Di Cardiologia Riabilitativa, Lumezzane, BS
  - Ospedale Monsignor Angelo R. Di Miccoli - Unita' Operativa Di Cardiologia, Barletta, BT
  - Ospedale Vittorio Emanuele Ii - Cardiologia, Bisceglie, BT
  - Azienda Ospedaliera G. Brotzu - Struttura Complessa Di Cardiologia, Cagliari, CA
  - Ospedale Ave Gratia Plena - Uosd Riabilitazione Cardiologica, San Felice A Cancello, CE
  - Ospedale San Giuseppe E Melorio U.O.C. Cardiologia Utic, Santa Maria Capua Vetere, CE
  - Ospedale S. Anna - U.O.C. Di Cardiologia, San Fermo della Battaglia, CO
  - Ospedale Maggiore - U.O. Cardiologia E Utic, Crema, CR
  - Ospedale Di Cremona - Uo Di Cardiologia, Cremona, CR
  - P.O. Garibaldi-Nesima - U.O.C. Di Cardiologia, Catania, CT
  - P.O. Garibaldi Centro - U.O.C. Cardiologia, Catania, CT
  - Policlinico Catania Po G. Rodolico - Ssd Scompenso Cardiaco Grave, Catania, CT
  - Ospedale Giovanni Paolo Ii - U.O. Cardiologia E Utic, Lamezia Terme, CZ
  - Ospedale M.Bufalini - U.O. Di Cardiologia-Utic, Cesena, FC
  - Ospedale G.B. Morgagni - L. Pierantoni - U.O. Cardiologia, Forlì, FC
  - Arcispedale Sant'Anna - U.O. Cardiologia - Utic, Ferrara, FE
  - Ospedali Riuniti - S.C. Di Cardiologia Univ.-Utic, Foggia, FG
  - Ospedale Civile San Giuseppe - Cardiologia, Empoli, FI
  - Ospedale Santa Maria Nuova - Hdu Cardiologica/Utic, Florence, FI
  - Ospedale San Giovanni Di Dio - Cardiologia, Florence, FI
  - Aou Careggi - Geriatria - Utig, Florence, FI
  - Ospedale Civile Augusto Murri - U.O. Cardiologia, Fermo, FM
  - Ospedale Policlinico San Martino - Unita' Operativa Cardiologia, Genova, GE
  - Ospedale Villa Scassi - Sc Cardiologia Utic, Genova, GE
  - Ospedale Padre Antero Micone - Sc Cardiologia - Utic, Genova, GE
  - Ospedale San Leopoldo Mandic - Cardiologia - Ucc, Merate, LC
  - Ospedale San Giuseppe Da Copertino - U.O. Di Cardiologia-Utic, Copertino, LE
  - Nuovo Ospedale Versilia - Sc Cardiologia, Lido di Camaiore, LU
  - Ospedale San Gerardo - U.O. Cardiologia-Utic, Monza, MB
  - Policlinico Di Monza - Uo Cardiol. Clinica E Scompenso Cardiaco, Monza, MB
  - Policlinico G. Martino - U.O. Medicina Interna, Messina, ME
  - Ospedale Civile - Uo Cardiologia, Legnano, MI
  - Ospedale San Raffaele - Cardiologia Clinica, Milan, MI
  - Centro Cardiologico Monzino - Cardiologia D'Urgenza, Milan, MI
  - Ospedale San Carlo Borromeo - Cardiologia-Ucc, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Diagnosi E Cure Terr. Malattie Cardiache, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 1 - Emodinamica, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 2 -Insuff. Card. E Trapianto, Milan, MI
  - Presidio Ospedaliero Di Passirana - Uo Cardiologia Riabilitativa, Rho, MI
  - Istituto Clinico Humanitas - U.O. Cardiologia Clinica, Rozzano, MI
  - Ospedale Ramazzini - U.O. Cardiologia, Carpi, MO
  - Ospedale Di Sassuolo - Cardiologia, Sassuolo, MO
  - Ospedale San Francesco - Cardiologia - Utic, Nuoro, NU
  - Fondazione G. Giglio - U.O. Cardiologia E Utic, Cefalù, PA
  - Ospedale Civile Immacolata Concezione - Cardiologia E Utic, Piove di Sacco, PD
  - Ospedale Di Assisi - Unita' Integrata Scompenso Cardiaco, Assisi, PG
  - Presidio Ospedaliero Citta' Di Castello - U.O. Di Cardiologia, Città di Castello, PG
  - Ex Ospedale Grocco - Unita' Operativa Cres, Perugia, PG
  - Azienda Ospedaliera Di Perugia - Cardiologia E Fisiopat. Cardiovascolare, Perugia, PG
  - Ftgm - Stabilimento Di Pisa - Cardiologia E Medicina Cardiovascolare, Pisa, PI
  - Ospedale Di Pordenone - S.O.C. Cardiologia, Pordenone, PN
  - Ics Maugeri Spa Societa' Benefit - Divisione Di Cardiologia Riabilitativa, Montescano, PV
  - Fondazione Irccs Policlinico San Matteo - Cardiologia, Pavia, PV
  - Ics Maugeri Spa Societa' Benefit - U.O. Di Riabilitazione Cardiologica, Pavia, PV
  - Ospedale Civile Santa Maria Delle Croci - U.O. Di Cardiologia, Ravenna, RA
  - Ospedale Civile San Sebastiano - Sos Cardiologia Area Nord, Correggio, RE
  - Ospedale Civile - Sc Cardiologia Area Nord, Guastalla, RE
  - Arcispedale Santa Maria Nuova - S.C. Cardiologia, Reggio Emilia, RE
  - Ospedale M.P. Arezzo - U.O.C. Cardiologia-Utic, Ragusa, RG
  - Aslrm6-Polo H2 Albano-Genzano - U.O.C. Di Cardiologia E Utic, Albano Laziale, RM
  - Ospedali Riuniti Anzio-Nettuno - U.O. Di Cardiologia - Utic, Anzio, RM
  - Policlinico Citta' Di Pomezia S. Anna - U.O. Cardiologia-Utic, Pomezia, RM
  - P.O. San Filippo Neri - Asl Roma 1 - Uoc Cardiologia E Utic, Roma, RM
  - Clinica Citta' Di Roma - Cardiologia-Utic, Roma, RM
  - Ospedale San Camillo - Uoc Cardiologia 1, Roma, RM
  - Policlinico Umberto Primo - Malattie Cardiovascolari A, Roma, RM
  - Policlinico Casilino - U.O. Cardiologia, Roma, RM
  - Ao San Giovanni Addolorata - Cardiologia E Riab. Cardiologica, Roma, RM
  - Ospedale Santo Spirito - U.O.C. Di Cardiologia, Roma, RM
  - Ospedale G. Ceccarini - Cardiologia-Utic, Riccione, RN
  - Ospedale Infermi -U.O. Cardiologia, Rimini, RN
  - Presidio Osped. S. Maria Della Speranza - U.O. Di Cardiologia, Battipaglia, SA
  - Ospedale Maria Ss. Addolorata - U.O. Di Cardiologia Utic, Eboli, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Cardiologia Interventistica - Emodinamic, Salerno, SA
  - Ospedale Dell'Alta Val D'Elsa Uosd Cardiologia-Utic, Poggibonsi, SI
  - Aou Senese Ospedale S. Maria Alle Scotte - U.O.C. Cardiologia Ospedaliera, Siena, SI
  - Ospedale E. Muscatello - U.O. Di Cardiologia - Utic, Augusta, SR
  - Ospedale G. Di Maria - Cardiologia Utic, Avola, SR
  - P.O. Lentini - U.O. Di Cardiologia Con Utic, Lentini, SR
  - Ospedale Civile G. Mazzini - Cardiologia Utic Ed Emodinamica, Teramo, TE
  - Por Cirie'- Lanzo Presidio Cirie' - S.C. Cardiologia Cirie'- Ivrea, Cirié, TO
  - Ospedale Civile - S.C. Cardiologia Cirie' Ivrea, Ivrea, TO
  - Ospedale Santa Croce - Cardiologia, Moncalieri, TO
  - Ospedale San Luigi Gonzaga - S.C.D.O. Cardiologia, Orbassano, TO
  - Ospedale Mauriziano Umberto I - Sc Cardiologia, Torino, TO
  - Maria Pia Hospital - Uo Medicina, Torino, TO
  - Ospedale Giovanni Bosco - Sc Cardiologia, Torino, TO
  - Asui Trieste - S.C. Centro Cardiovascolare, Trieste, TS
  - Ospedali Riuniti - Osp. Cattinara - S.O.C. Cardiologia, Trieste, TS
  - Ospedale Ca' Foncello - U.O.C. Cardiologia, Treviso, TV
  - Pou Santa Maria Della Misericordia - S.O.C. Cardiologia, Udine, UD
  - Ospedale Di Circolo Di Busto Arsizio - Uoc Cardiologia Utic Emodinamica, Busto Arsizio, VA
  - Ospedale S. Antonio Abate - U.O. Di Cardiologia, Gallarate, VA
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale Di Circolo E Fondazione Macchi - Cardiologia I, Varese, VA
  - Ospedale Civile - U.O.C. Cardiologia, Chioggia, VE
  - Ospedale Civile - U.O. Cardiologia, Mirano, VE
  - Ospedale Civile - U.O.C. Cardiologia, Arzignano, VI
  - Ospedale G. Fracastoro - U.O.C. Di Cardiologia, San Bonifacio, VR
  - Ospedale Civile G. Jazzolino - U.O. Cardiologia - Utic, Vibo Valentia, VV
  - Ospedale San Giovanni Di Dio - Uo Cardiologia - Utic, Frattamaggiore
  - Ospedale Generale Di Zona - U.O. Cardiologia - Utic, Giugliano in Campania
  - Aou Federico Ii - Uoc Cardiologia E Utic, Napoli
  - Pres. Ospedaliero S. Maria Della Pieta' - U.O. Cardiologia E Utic, Nola
  - Ospedale Della Val Di Nievole - U. O. Cardiologia - Utic, Pescia
  - Ospedale San Jacopo - U.O. Cardiologia, Pistoia
  - Casa Di Salute Santa Lucia - U.O. Cardiologia, San Giuseppe Vesuviano